CLINICAL TRIAL: NCT04177498
Title: A Pilot, Open Study to Assess Efficacy and Safety of Rigosertib in Patients With Recessive Dystrophic Epidermolysis Bullosa Associated Locally Advanced/Metastatic Squamous Cell Carcinoma
Brief Title: Rigosertib in Patients With Recessive Dystrophic Epidermolysis Bullosa Associated SCC
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: Traws Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19G.527; JT 13813 (Other: JeffTrial Number)
Record Dates: First submitted 2019-11-07; First posted 2019-11-26 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Recessive Dystrophic Epidermolysis Bullosa
MeSH Terms: conditions — Epidermolysis Bullosa Dystrophica | interventions — ON 01910

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (rigosertib sodium) (Experimental): Patients receive rigosertib sodium either oral or IV over a 52 week period. Patients will take oral rigosertib continuously for a total of three weeks, every four-week cycle (three weeks on, one week off drug). For IV, rigosertib is administered as a 72-hr continuous infusion on Days 1, 2 and 3 of a 2-week cycle for the first eight 2-week cycles, then on Days 1, 2 and 3 of a 4-week cycle thereafter.
  Interventions: Drug: Rigosertib Sodium; Other: Quality-of-Life Assessment

INTERVENTIONS:
Drug: Rigosertib Sodium — given PO or 72 hour continuous infusion
  Other Names: ON 01910.Na
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This pilot trial studies how rigsertib sodium works in treating patients with Recessive Dystrophic Epidermolysis bullosa (RDEB) with locally advanced Squamous Cell Carcinoma (SCC). Rigosertib may selectively target Epidermolysis bullosa (EB) cancer cells while leaving normal EB cells unaffected.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the anti-tumor activity of oral or IV rigosertib in RDEB patients with advanced SCC that have failed prior standard of care, by determining the overall response rate (ORR) which is defined as the proportion of patients who achieve either a CR or a PR by RECIST v1.1 II. To evaluate the safety and tolerability of oral rigosertib administered either orally daily three weeks on, one week off or as 72h CIV infusions on day 1-3 of a two week-cycle for 8 cycles and then on day 1-3 of a 4 week cycle thereafter

SECONDARY OBJECTIVES:

I. Assess impact on quality of life (QoL) II. Biomarker analysis (to include markers of PI3K/Akt and PLK1 pathways) performed on all archival tissue from all patients

EXPLORATORY OBJECTIVE:

I. Exome sequencing of patient tumors before, during, and after treatment

OUTLINE: Patients will receive rigosertib sodium as either oral capsules or IV infusion. Mode of application is determined by the responsible investigator depending on participant's needs, general condition, and possibility of ambulatory treatment or need of hospitalization.

Patients will take oral rigosertib continuously for a total of three weeks of a four-week cycle (three weeks on, one week off drug).

For IV treatment, patients will receive rigosertib IV administered as a 72-hr continuous infusion on Days 1, 2 and 3 of a 2-week cycle for the first eight 2-week cycles, then on Days 1, 2 and 3 of a 4-week cycle thereafter.

Patients will receive treatment over a 52 week period. After completion of study treatment, patients are followed periodically every 3 months over a 12 month period.

ELIGIBILITY:
Inclusion Criteria:

1. 18-79 years of age;
2. Diagnosis of RDEB associated unresectable, locally advanced or metastatic SCC of the skin confirmed prior to the Screening Visit.
3. Failure to respond to SCC standard of care as follows; surgical excision, radiotherapy and conventional chemotherapy with e.g. platin derivates (i.e., cisplatin carboplatin) or cetuximab, 5-fluorouracil, bleomycin, methotrexate, adriamycin, taxanes, gemcitabine or ifosfamide alone or in combination; or failure to respond to previous alternative biologic treatments such as epidermal growth factor inhibitors (like cetuximab and panitumumab) or immune checkpoint (programmed cell death 1) inhibitors (such as nivolumab, pembrolizumab, cempilimab). For recent guidelines on standard of care for RDEB SCC and non EB-SCC
4. Is not currently receiving any other cancer therapy.
5. Measurable disease based on Response Criteria in Solid Tumors Version 1.1 (RECIST 1.1)
6. Patient (or patient's legally authorized representative) must have signed an informed consent document indicating that the patient understands the purpose of and procedures required for the study and is willing to participate in the study.

Exclusion Criteria:

1. Response to standard of care a. Surgical excision, radiotherapy and or conventional chemotherapy with e.g. platin derivates (i.e., cisplatin, carboplatin) or cetuximab, 5-fluorouracil, bleomycin, methotrexate, adriamycin, taxanes, gemcitabine or ifosfamide alone or in combination; or alternative biologic treatments such as epidermal growth factor inhibitors (like cetuximab and panitumumab) or immune checkpoint (programmed cell death 1) inhibitors (such as nivolumab, pembrolizumab, cempilimab). For recent guidelines on standard of care for RDEB SCC and non EB-SCC
2. Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure or unstable angina pectoris
3. Active systemic infection not adequately responding to appropriate therapy
4. Total bilirubin ≥ 1.5 mg/dL not related to hemolysis or Gilbert's disease, ≥5.3 mg/dL in patients if related to hemolysis or Gilbert's disease
5. Alanine transaminase (ALT)/aspartate transaminase (AST) ≥ 2.5 x upper limit of normal (ULN)
6. Serum creatinine ≥2 .0 mg/dL or eGFR (estimated Glomerular Filtration Rate) <60 mL/min.
7. White blood cell count ≤ 2000/μl OR Neutrophils ≤ 1500/μL OR Platelets ≤ 100 x103/μL OR Hemoglobin ≤ 7.9 g/dL
8. Known active HIV, hepatitis B or hepatitis C, where active is defined as follows: a. HIV or Hepatitis C - presence of viral load b. Hepatitis B - antigen positive
9. Uncorrected hyponatremia (defined as serum sodium value of <125 mmol/L)
10. Female patients of child-bearing potential and male patients with partners of childbearing potential who are unwilling to follow strict contraception requirements throughout the study, up to and including the 30-day non-treatment follow-up period
11. Female subjects: pregnant or lactating women and all women physiologically capable of becoming pregnant (i.e. women of childbearing potential) UNLESS they are willing to use one or more reliable methods of contraception with a Pearl index ≤1 including combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (either oral or intravaginal or transdermal); progestogen-only hormonal contraception associated with inhibition of ovulation (either oral or injectable or implantable); an intrauterine device (IUD); an intrauterine hormone-releasing system ( IUS); bilateral tubal occlusion; vasectomised partner or sexual abstinence. Reliable contraception should be maintained throughout the study. A pregnancy test in urine will be performed at screening in all women of childbearing potential, and repeated before biopsy treatment and at all visits. Any postmenopausal women (physiologic menopause defined as "12 consecutive months of amenorrhea") or women permanently sterilized (e.g. tubal occlusion, hysterectomy or bilateral salpingectomy) will not be required to undergo pregnancy test.
12. Uncontrolled hypertension a. (i.e. systolic blood pressure greater than or equal to 140mmHg and diastolic blood pressure greater than or equal to 90mmHg despite intake of ≥ 3 antihypertensive medications with complementary mechanisms of action (a diuretic should be 1 component)
13. Patient is currently participating and receiving study therapy or systemic therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
14. Psychiatric illness or social situation that would limit the patient's ability to tolerate and/or comply with study requirements
15. Patients (or patient's legally authorized representative) unlikely to comply with the study protocol or unable to understand the nature and scope of the study or the possible benefits or unwanted effects of the study procedures and treatments.
16. History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the patient to participate, in the opinion of the treating Investigator
17. Known hypersensitivity reaction to any of the components of study treatment
18. Any patient with a known medical condition leading to abnormal vital signs that is not correctable or a patient whose vital sign is within abnormal range upon arrival in clinic will not be receiving the medication. If this abnormal vital signs are not medically controlled and addressed that patient will be excluded at anytime (regardless of it is at arrival or in the middle of the study).

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-08-24 (Actual); Primary Completion 2025-05-05 (Actual); Study Completion 2025-05-05 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | baseline up to12 months post treatment
  Defined as the proportion of patients who achieve either a complete response (CR) or partial response (PR)
Incidence of treatment-related adverse events | baseline up to12 months post treatment
  Safety assessments will be based on medical review of adverse event reports and the results of vital sign measurements, physical examinations, and clinical laboratory tests. Results will be reported as an aggregate of the adverse events using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), Version 5.0 terminology and grading.

SECONDARY OUTCOMES:
Quality of Life Epidermolysis Bullosa (QOLEB) questionnaire | baseline up to12 months post treatment
  Descriptive methods used to analyze scores from QOLEB questionnaire. It consists of 17 questions with four response choices from "not at all" to "constant"
Biomarker Analysis | baseline up to12 months post treatment
  Fixed tissue will be assessed using immuno-histochemistry with antibodies raised against phosphorylated AKT (p473 Akt), phosphorylated C-RAF (p-S338 RAF), phosphorylated ERK and cleaved caspase.
Efficacy of rigosertib sodium treatment: The Objective Response Rate | baseline to end of treatment (52 weeks)
  The Objective Response Rate (ORR) will be computed with the corresponding exact binomial 90% confidence interval.

OTHER OUTCOMES:
Exosome sequencing | baseline up to12 months post treatment
  whole exosome sequencing will be done on frozen tumor tissue. The investigators will catalogue somatic mutations identified in each tumor and compare these data with patient response and ex-vivo tumor responses.

CONTACTS AND LOCATIONS:
Overall Officials: Neda Nikbakht, MD, PhD, Principal Investigator — Sidney Kimmel Cancer Center at Thomas Jefferson University
Locations (1):
- Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No